CLINICAL TRIAL: NCT01363076
Title: A Study of the Pharmacokinetics of Ketorolac Tromethamine Administered Intranasally (IN) for Postoperative Pain in Children Aged 12 Through 17 Years
Brief Title: The Pharmacokinetics of Ketorolac Tromethamine Administered Intranasally (IN) for Postoperative Pain in Children Aged 12 Through 17 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROX 2006-02
Record Dates: First submitted 2011-05-27; First posted 2011-06-01 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac Tromethamine

ARMS (2):
- Ketorolac Tromethamine (15 mg) (Experimental): Ketorolac Tromethamine - single dose (15 mg) administered intranasally (IN) for subjects weighing <50 kg.
  Interventions: Drug: Ketorolac Tromethamine
- Ketorolac Tromethamine (30 mg) (Experimental): Ketorolac Tromethamine - single dose (30 mg) administered intranasally (IN) for subjects weighing ≥50 kg.
  Interventions: Drug: Ketorolac Tromethamine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Single IN dose of 15 mg ketorolac tromethamine for subjects weighing <50 kg.
  Arms: Ketorolac Tromethamine (15 mg)
Drug: Ketorolac Tromethamine — Single IN dose of 30 mg ketorolac tromethamine for subjects weighing ≥50 kg.
  Arms: Ketorolac Tromethamine (30 mg)

SUMMARY:
This was an open-label PK study in pediatric subjects who had undergone general surgery. Each subject's study participation consisted of a screening visit, a single-dose treatment with intranasal ketorolac (IN) tromethamine, and a follow-up visit.

Following surgery, subjects received IN ketorolac 15 mg (weight < 50 kg) or 30 mg (weight > or = 50 kg) when pain relief was indicated. For pain not relieved by the study drug, the subjects had access to an opioid analgesic administered by patient-controlled analgesia (PCA). Blood samples for pharmacokinetic analysis were obtained at specified time points following the dose of ketorolac.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12 through 17 years
* Body weight > or = 30 kg and < or = 100 kg
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test result prior to entry into the study
* A legal representative able to provide written informed consent
* Willing and able to comply with all testing and requirements defined in the protocol
* Willing and able to complete the posttreatment visit

Exclusion Criteria:

* Allergy or sensitivity to ketorolac or ethylene diamine tetraacetic acid (EDTA)
* Allergic reaction to aspirin or other NSAIDs
* Had an upper respiratory tract infection or other respiratory tract condition (eg, active allergic rhinitis) that could interfere with the absorption of the nasal spray or with the assessment of AEs
* Use of any IN product within 24 hours prior to study entry
* Clinically significant abnormality on screening laboratory tests
* History of cocaine use resulting in nasal mucosal damage
* History of peptic ulcer disease or gastrointestinal bleeding
* Had advanced renal impairment or a risk for renal failure due to volume depletion
* A history of any other clinically significant medical problem, which in the opinion of the investigator would interfere with study participation
* Participation within 30 days of study entry or within 5 times the half-life, whichever is longer, in another investigational drug study
* Allergy or significant reaction to opioids
* Was pregnant or breastfeeding
* Previously participated in this study
* The surgical procedure involved head, neck, oral, or nasal surgery

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln Bynum, MD, Study Chair — ICON Developmental Solutions
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 2007 - January 2008; Location: Stanford University Medical Center
Pre-assignment Details: Screening procedure consisting of an interview and the following assessments: demographics, medical history, physical examination, concomitant medications within last 30 days, vital signs, clinical laboratory tests, pregnancy test (female subjects).
Groups:
- Ketorolac Tromethamine (15 mg): Single intranasal (IN) dose of 15 mg ketorolac tromethamine for subjects weighing <50 kg.
- Ketorolac Tromethamine (30 mg): Single intranasal (IN) dose of 30 mg ketorolac tromethamine for subjects weighing ≥50 kg.
Period: Overall Study
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Started | 7 | 13
Completed | 7 | 12
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg) | Total
Number analyzed (Participants) | 7 | 13 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 13 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.1 (0.7) | 15.4 (1.6) | 15.0 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 4 | 9 | 13
Region of Enrollment [Number; unit: participants]
  United States | 7 | 13 | 20

OUTCOME MEASURES:

1. Primary Outcome: Cmax (the Maximum Observed Plasma Concentration)
Description: Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Professional. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each dose level, together with the individual plasma concentrations of ketorolac.
Time Frame: All PK parameters were assessed using blood samples collected 15 minutes prior to the dose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, 8, 12, and 24 hours after the dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Number analyzed (Participants) | 7 | 13
ng/mL | 1153.9 (485.0) | 1625.3 (538.5)

2. Primary Outcome: Tmax (The Time to Maximum Observed Plasma Concentration; ie. The Time at Which Cmax Occured)
Description: Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Pro. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each dose level, together with the individual plasma concentrations of ketorolac. Individual plasma ketorolac concentrations were summarized by dose level for the PK population at each sampling time using n, arithmetic mean, SD, CV(%), geometric mean, 95% confidence intervals (CI) for the arithmetic mean, median, minimum, and maximum.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Number analyzed (Participants) | 7 | 13
hr | 0.720 [0.38 to 6.07] | 0.780 [0.48 to 5.00]

3. Primary Outcome: AUClast (the Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Last Quantifiable Timepoint Post-dose)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Number analyzed (Participants) | 7 | 13
ng•h/mL | 9308.2 (6214.2) | 10662.1 (5383.5)

4. Primary Outcome: AUCinf (the AUC Time From Zero to Infinity, Where Possible)
Description: Pharmacokinetic analysis by standard model independent methods was performed by a pharmacokineticist using WinNonlin Pro. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each dose level, together with the individual plasma concentrations of ketorolac. AUCinf calculated as: AUCinf = AUC(0-24) + (concentration at 24 hr/elimination constant).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Number analyzed (Participants) | 6 | 12
ng•h/mL | 10590.7 (7818.4) | 11949.5 (6506.1)

5. Primary Outcome: AUC 0-24 (the AUC From Time Zero to 24 Hours Post-dose
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng•h/mL
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Number analyzed (Participants) | 7 | 12
ng•h/mL | 9600.5 (5959.9) | 11317.2 (5666.1)

6. Primary Outcome: t1/2 (the Terminal Half-life, Where Possible)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Number analyzed (Participants) | 6 | 12
hr | 6.678 (2.882) | 5.031 (2.055)

7. Primary Outcome: MRT (Mean Residence Time)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Number analyzed (Participants) | 6 | 12
hr | 9.664 (3.892) | 6.727 (1.945)

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Ketorolac Tromethamine (15 mg) | Ketorolac Tromethamine (30 mg)
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/13
Other Adverse Events (participants affected / at risk) | 3/7 | 8/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac Tromethamine (15 mg) (N=7) | Ketorolac Tromethamine (30 mg) (N=13)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac Tromethamine (15 mg) (N=7) | Ketorolac Tromethamine (30 mg) (N=13)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No